CLINICAL TRIAL: NCT04049461
Title: The Causes of Heterotopic Ossification in Abdominal Incision After Pancreatic Surgery：A Single-center Prospective Study
Brief Title: Heterotopic Ossification in Abdominal Incision and Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yi Miao, Prof., Director of Pancreas Center, Nanjing Medical University
Other Study IDs: NMU-JSPH-PC-Ossification
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Cancer of Pancreas; Ossification, Heterotopic
Keywords: Cancer of Pancreas; Ossification, Heterotopic; Abdominal incision
MeSH Terms: conditions — Pancreatic Neoplasms; Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The ossification patients were sequenced with informed consent . Promise to keep their personal information confidential.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDAC Group: Radical operations were performed through central abdominal incisions. The postoperative pathology was pancreatic ductal adenocarcinoma.
  Interventions: Diagnostic Test: Bone alkaline phosphatase; Radiation: Abdominal CT scan
- Benign Group: The abdominal midline incision was performed and the postoperative pathology was benign.
  Interventions: Diagnostic Test: Bone alkaline phosphatase; Radiation: Abdominal CT scan

INTERVENTIONS:
Diagnostic Test: Bone alkaline phosphatase — Hematologic indicators reflecting ossification.
Radiation: Abdominal CT scan — Observe whether HOAI occurs.

SUMMARY:
To investigate whether pancreatic cancer is the cause of heterotopic ossification of abdominal incision.

DETAILED DESCRIPTION:
Heterotopic ossification of abdominal incision (HOAI) has long been regarded as a rare complication after general surgery. However,according to our retrospective analysis. HOAI was more frequently observed in the malignancy group (33/121 cases, 27.3%) than in the non- malignancy group. Because of the many biases in the retrospective analysis, the result was not widely shared.

The purpose of this prospective study is to confirm that pancreatic cancer is the cause of heterotopic ossification of abdominal incisions. According to postoperative pathology, the patients were divided into two groups: pancreatic cancer group and benign diseases group.The researchers will observe whether patients develop heterotopic ossification of the abdominal incision one year after surgery to conclude.

ELIGIBILITY:
Inclusion Criteria:

* Obtain informed consent from the patients.
* The patient's abdominal incision was double-closed with continuous suture of linea alba and fascia with absorbable suture, and skin was sutured with skin staples.

Exclusion Criteria:

* Refusing to join the study
* Previous history of malignant tumor
* Previous history of midabdominal incision
* Abnormal calcium and phosphorus metabolism
* Distant metastasis
* Palliative operation
* performing neoadjuvant chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Han population
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HOAI | 12 months
  HOAI is determined by CT, whose CT number is similar to that of the same spine.
Bone alkaline phosphatase | 12 months
  Preoperative tests were performed and every three months postoperatively

SECONDARY OUTCOMES:
Incidence of distant metastasis and local recurrence | 12 months
  Patients with pancreatic cancer were divided into HOAI and non-HOAI groups to determine whether there were differences in the incidence of distant metastasis and local recurrence between the two groups.

OTHER OUTCOMES:
Overall survival | 5 years
  Patients with pancreatic cancer were divided into HOAI and non-HOAI groups to determine whether there were differences between the OS of two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Miao, Prof., Principal Investigator — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University; Junli Wu, MD,PHD, Study Director — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University; Jishu Wei, MD,PHD, Principal Investigator — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Ghuman MS, Saggar K. Images in clinical medicine. Heterotopic ossification of a midline abdominal incision. N Engl J Med. 2014 Jul 31;371(5):464. doi: 10.1056/NEJMicm1312006. No abstract available. PMID 25075838
- [Background] Kim J, Kim Y, Jeong WK, Song SY, Cho OK. Heterotopic ossification developing in surgical incisions of the abdomen: analysis of its incidence and possible factors associated with its development. J Comput Assist Tomogr. 2008 Nov-Dec;32(6):872-6. doi: 10.1097/RCT.0b013e318159c617. PMID 19204446
- [Background] Koolen PG, Schreinemacher MH, Peppelenbosch AG. Heterotopic ossifications in midline abdominal scars: a critical review of the literature. Eur J Vasc Endovasc Surg. 2010 Aug;40(2):155-9. doi: 10.1016/j.ejvs.2010.03.010. Epub 2010 Apr 18. PMID 20400341
- [Background] Isaacson BM, Potter BK, Bloebaum RD, Epperson RT, Kawaguchi BS, Swanson TM, Pasquina PF. Link Between Clinical Predictors of Heterotopic Ossification and Histological Analysis in Combat-Injured Service Members. J Bone Joint Surg Am. 2016 Apr 20;98(8):647-57. doi: 10.2106/JBJS.15.00895. PMID 27098323
- [Background] Citak M, Grasmucke D, Suero EM, Cruciger O, Meindl R, Schildhauer TA, Aach M. The roles of serum alkaline and bone alkaline phosphatase levels in predicting heterotopic ossification following spinal cord injury. Spinal Cord. 2016 May;54(5):368-70. doi: 10.1038/sc.2015.211. Epub 2015 Dec 8. PMID 26643987